CLINICAL TRIAL: NCT01676701
Title: Pharmacokinetic Evaluations of Tabalumab Following Subcutaneous Administration by Prefilled Syringe or Auto Injector in Patients With Rheumatoid Arthritis Who Have Had an Inadequate Response to Methotrexate
Brief Title: Evaluation of Tabalumab Using Auto-Injector or Prefilled Syringe in Participants With Rheumatoid Arthritis (RA)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient efficacy observed in study BCDM(NCT01198002) and BCDV(NCT01202773)
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14598; H9B-MC-BCEF (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Results first posted 2018-04-26 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tabalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tabalumab Auto-Injector (Experimental): Tabalumab 180 milligram (mg) loading dose administered using auto-injectors at Week 0 as 2 subcutaneous (SC) injections (90 mg each), followed by a 90 mg SC injection every 2 weeks (Q2W) up to Week 12.
  Interventions: Drug: Tabalumab Auto-Injector
- Tabalumab Prefilled Syringe (Experimental): Tabalumab 180 mg loading dose administered using prefilled syringes at Week 0 as 2 SC injections (90 mg each), followed by a 90 mg SC injection Q2W up to Week 12.
  Interventions: Drug: Tabalumab Prefilled Syringe

INTERVENTIONS:
Drug: Tabalumab Auto-Injector — Administered SC by auto-injector
  Other Names: LY2127399
  Arms: Tabalumab Auto-Injector
Drug: Tabalumab Prefilled Syringe — Administered SC by prefilled syringe
  Other Names: LY2127399
  Arms: Tabalumab Prefilled Syringe

SUMMARY:
The purpose of this study is to evaluate the serum concentration of tabalumab after the administration using either prefilled syringe or auto-injector after the initial loading dose and after 12 weeks of treatment. Treatment period is followed by 40 weeks optional safety extension.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory males or females ≥18 years of age
* Diagnosis of adult-onset RA
* Active RA (at least 8/68 tender and at least 8/66 swollen joints)
* Screening C-reactive protein (CRP) >1.2 times the upper limit of normal (ULN) or a screening erythrocyte sedimentation rate (ESR) >28 millimeters per hour (mm/hr)
* Documented history of, or current, positive rheumatoid factor (RF) and/or anti-cyclic citrullinated peptide antibody (anti-CCP Ab) test
* Regular use of methotrexate (MTX) for at least 12 weeks and stable dose (10 to 25 mg/week) for at least 8 weeks prior to baseline
* American College of Rheumatology (ACR) functional class I, II, or III
* Able and willing to inject tabalumab by themselves (or have an assistant who will inject tabalumab) and able and willing to complete all study procedures
* Able and willing to have blood drawn for pharmacokinetic (PK) sampling

Exclusion Criteria:

* Use of oral corticosteroids at average daily doses of >10 milligrams per day (mg/day) of prednisone or its equivalent within 6 weeks prior to baseline
* Injection of any parenteral (including intraarticular) corticosteroid within 6 weeks of baseline
* Have previously discontinued treatment with a biologic disease-modifying antirheumatic drug (DMARD) or a novel drug that interrupts cytokine signaling [for example, Janus kinase (JAK) inhibitors] due to insufficient efficacy
* Participants who had discontinued biologic DMARDS for reasons other than efficacy will not be excluded but must have done so prior to baseline
* Participants who discontinued a JAK inhibitor for lack of efficacy
* Participants who discontinued a JAK inhibitor for reasons other than efficacy will not be excluded, but must have done so prior to baseline for 21 days
* Previous severe reaction to any biologic therapy that, in the opinion of the Investigator, would pose an unacceptable risk to the participant if participating in the study
* Have had an inadequate response to treatment with 3 or more of the following DMARDs prescribed alone or in combination at approved doses for a minimum of 90 days: leflunomide, azathioprine, cyclosporine, and/or sulfasalazine
* Use of other DMARDs (for example, gold salts, cyclosporin, azathioprine, or any other immunosuppressives) other than MTX, hydroxychloroquine, chloroquine, or sulfasalazine, or the use of a JAK inhibitor in the 8 weeks prior to baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (37):
- United States (14):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glendale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lewes, Delaware
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., DeBary, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tamarac, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prairie Village, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lansing, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Freehold, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wyomissing, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
- Argentina (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Córdoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Quilmes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Miguel de Tucumán
- Czechia (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hostivice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plzen-Bory
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Uherské Hradiště
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zlín
- Poland (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bydgoszcz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elblag
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
- Puerto Rico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponce
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santurce
- Russia (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saratov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulyanovsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yaroslavl

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was to include a 12-week treatment period, optional 40-week safety extension, and post-treatment follow-up (at least 24 weeks). At the time of early study termination, all participants who had received tabalumab discontinued dosing and then completed the post-treatment follow-up period. No one entered the 40-week safety extension period.
Groups:
- Tabalumab Auto-Injector: Tabalumab: Using auto-injectors, participants received a 180 milligram (mg) loading dose at Week 0 as 2 subcutaneous (SC) injections (90 mg each). Participants also received a 90 mg SC injection every 2 weeks (Q2W) until early study termination (up to Week 6).
- Tabalumab Prefilled Syringe: Tabalumab: Using prefilled syringes, participants received a 180 mg loading dose administered at Week 0 as 2 SC injections (90 mg each). Participants also received a 90 mg SC injection Q2W until early study termination (up to Week 6).
Period: Overall Study
Arm/Group | Tabalumab Auto-Injector | Tabalumab Prefilled Syringe
Started | 4 | 4
Received at Least 1 Dose of Study Drug | 4 | 4
Completed Post-Treatment Follow-Up | 4 | 4
Completed | 0 | 0
Not Completed | 4 | 4
Not completed — Protocol Violation | 1 | 0
Not completed — Sponsor Decision | 3 | 4

BASELINE CHARACTERISTICS:
Population: Randomized participants who received at least 1 dose of study drug.
Groups:
- Tabalumab Auto-Injector: Tabalumab: Using auto-injectors, participants received a 180 mg loading dose administered at Week 0 as 2 SC injections (90 mg each). Participants also received a 90 mg SC injection Q2W until early study termination (up to Week 6).
- Total: Total of all reporting groups
Arm/Group | Tabalumab Auto-Injector | Tabalumab Prefilled Syringe | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Customized [Number; unit: participants]
  43.3 to 65.4 years | 4 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Serum Concentration (Cmax) of Tabalumab After Loading Dose
Time Frame: Days 4, 7, 9, 11, and 14 after loading dose administered
Population: No participant had outcome measure data analyzed due to the termination of the trial and an insufficient sample size.
Arm/Group | Tabalumab Auto-Injector | Tabalumab Prefilled Syringe
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: PK: Area Under the Concentration Time Curve From Time 0 to 14 Days [AUC(0-14)]
Time Frame: Days 4, 7, 9, 11, and 14 after loading dose administered
Population: No participant had outcome measure data analyzed due to the termination of the trial and an insufficient sample size.
Arm/Group | Tabalumab Auto-Injector | Tabalumab Prefilled Syringe
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline to 12-Week Endpoint in Achieving American College of Rheumatology (ACR) Core Set
Time Frame: Baseline, Week 12
Population: No participant had outcome measure data analyzed due to the termination of the trial and an insufficient sample size.
Arm/Group | Tabalumab Auto-Injector | Tabalumab Prefilled Syringe
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Participants Achieving ACR Response
Time Frame: Week 12
Population: No participant had outcome measure data analyzed due to the termination of the trial and an insufficient sample size.
Arm/Group | Tabalumab Auto-Injector | Tabalumab Prefilled Syringe
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percent Change From Baseline to 12-Week Endpoint in American College of Rheumatology (ACR-N) Index
Time Frame: Baseline, Week 12
Population: No participant had outcome measure data analyzed due to the termination of the trial and an insufficient sample size.
Arm/Group | Tabalumab Auto-Injector | Tabalumab Prefilled Syringe
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline to 12-Week Endpoint in Disease Activity Score Based on a 28-Joint Count and C-Reactive Protein (DAS28-CRP) Level
Time Frame: Baseline, Week 12
Population: No participant had outcome measure data analyzed due to the termination of the trial and an insufficient sample size.
Arm/Group | Tabalumab Auto-Injector | Tabalumab Prefilled Syringe
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percentage of Participants Achieving European League Against Rheumatism Responder Index Based on the 28-Joint Count (EULAR-28)
Time Frame: Week 12
Population: No participant had outcome measure data analyzed due to the termination of the trial and an insufficient sample size.
Arm/Group | Tabalumab Auto-Injector | Tabalumab Prefilled Syringe
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants Developing Anti-Tabalumab Antibodies
Time Frame: Week 12
Population: No participant had outcome measure data analyzed due to the termination of the trial and an insufficient sample size.
Arm/Group | Tabalumab Auto-Injector | Tabalumab Prefilled Syringe
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Operation Failures
Time Frame: Week 12
Population: No participant had outcome measure data analyzed due to the termination of the trial and an insufficient sample size.
Arm/Group | Tabalumab Auto-Injector | Tabalumab Prefilled Syringe
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline Score in Subcutaneous Administration Assessment Questionnaire (SQAAQ)
Time Frame: Baseline, Weeks 4 and 8
Population: No participant had outcome measure data analyzed due to the termination of the trial and an insufficient sample size.
Arm/Group | Tabalumab Auto-Injector | Tabalumab Prefilled Syringe
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 12 or early termination (Treatment Period) and last dose up to 24 weeks post last dose (Post-Treatment Follow-Up Period)
Groups:
- Tabalumab Auto-Injector (Treatment Period): Tabalumab: Using auto-injectors, participants received a 180 mg loading dose administered at Week 0 as 2 SC injections (90 mg each). Participants also received a 90 mg SC injection Q2W until early study termination (up to Week 6).
- Tabalumab Auto-Injector (Post Treatment Follow-Up Period): No study drug was administered during the Post-Treatment Follow-Up Period for participants in the Tabalumab Auto-Injector treatment arm.
- Tabalumab Prefilled Syringe (Treatment Period): Tabalumab: Using prefilled syringes, participants received a 180 mg loading dose administered at Week 0 as 2 SC injections (90 mg each). Participants also received a 90 mg SC injection Q2W until early study termination (up to Week 6).
- Tabalumab Prefilled Syringe (Post Treatment Follow-Up Period): No study drug was administered during the Post-Treatment Follow-Up Period for participants in the Tabalumab Prefilled Syringe treatment arm.
Arm/Group | Tabalumab Auto-Injector (Treatment Period) | Tabalumab Auto-Injector (Post Treatment Follow-Up Period) | Tabalumab Prefilled Syringe (Treatment Period) | Tabalumab Prefilled Syringe (Post Treatment Follow-Up Period)
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 1/4 | 0/4 | 0/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tabalumab Auto-Injector (Treatment Period) (N=4) | Tabalumab Auto-Injector (Post Treatment Follow-Up Period) (N=4) | Tabalumab Prefilled Syringe (Treatment Period) (N=4) | Tabalumab Prefilled Syringe (Post Treatment Follow-Up Period) (N=4)
Gastric Infection (Infections and infestations) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to early termination of the trial, no participant had outcome measure data analyzed. Participants who received study treatment had disposition, demographic, and adverse event data reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days